CLINICAL TRIAL: NCT07009080
Title: Motor Imagery is Effective in the Prevention of Landing Errors in Volleyball Players: a Randomized Controlled Trial
Brief Title: The Effect of Motor Imagery on Preventing Volleyball Players During Jumping and Landing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydan Niziplioğlu (Other)
Responsible Party: Sponsor-Investigator, Aydan Niziplioğlu, MSc.Physiotherapist, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sportsMI
Record Dates: First submitted 2025-05-27; First posted 2025-06-06 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Motor Imagery
Keywords: prevention; motor imagery; volleyball; sports medicine

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- solo training (Experimental): Prior to the study, a video recording with the correct jump and landing kinematics, showing the correct hip, knee, and ankle flexion angles , will be recorded by the researchers. The video will be a minute long, consisting of front and side angles, and featured a professional volleyball player who won't be included in the study. Players in solo training group individually underwent the training.For standardization purposes, no questions will allowed during the training session. In the training session, players will be asked to watch the correct landing video at a slightly slower speed and contemplate the appropriate hip, knee, and ankle angles. Then, the researcher explained correct landing mechanics, while referring to the correct landing video, pointed out the common errors, and described how to correct them.The researcher then will explain to the players what MI is and how it works.
  Interventions: Other: motor imagery
- group training (Experimental): Prior to the study, a video recording with the correct jump and landing kinematics, showing the correct hip, knee, and ankle flexion angles, will be recorded by the researchers. The video will be a minute long, consisting of front and side angles, and featured a professional volleyball player who will not included in the study. Players in the GT group underwent the training as a group in a quiet, climate-controlled room. For standardization purposes, no questions were allowed during the training session. In the training session, players were asked to watch the correct landing video at a slightly slower speed and contemplate the appropriate hip, knee, and ankle angles. Then, the researcher explained correct landing mechanics, while referring to the correct landing video, pointed out the common errors, and described how to correct them.The researcher then will explain to the players what MI is and how it works.
  Interventions: Other: motor imagery
- control training (No Intervention): Players only participate in evaluations

INTERVENTIONS:
Other: motor imagery — The researcher will explain to the players what MI is and how it works. Following the explanation, players will seated in a comfortable armchair facing the researcher, will ask to minimize distracting thoughts, and to be as mindful as possible without speaking for five minutes, and to imagine themselves executing the correct angles during a landing.
  Arms: group training; solo training

SUMMARY:
Although the effectiveness of motor imagery in improving performance in sports is known, there is no research on its preventive role against injuries. the primary aim of this study is to investigate the effect of motor imagery on improving risk factors related to jumps and falls in volleyball players. The secondary aim of this study is to investigate the effect of motor imagery on cortical functions.

DETAILED DESCRIPTION:
The nature of volleyball includes serving, blocking, and/or spiking, which require players to jump frequently. This high demand on the lower extremity causes high injury rates: approximately 58.7% of all injuries involve lower extremities, among which 51.8% are non-contact injuries . The knee accounts for 58% of lower extremity injuries -15.2% of which involve ACL- while 25.9% affect the ankle, including ligament injuries, sprains, and strains . These high injury rates cause players to lose game-time, 4.49 per 1000 hours for competition and 3.43 per 1000 hours for practice hours and cause their clubs to lose money .

Most studies in the literature focused on ACL injuries and they reported numerous risk factors, such as anatomic, hormonal, biomechanical, and unanticipated. Of these biomechanical risk factors, increased anterior tibial shear force, decreased knee flexion while landing, increased knee valgus, knee and hip internal rotation, and hip adduction were reported as the most important. These joint angle errors are reported to be the cause of 47.5% of the knee injuries in volleyball during jumping and falling . Also, altered kinetics in landing are suggested to potentially increase risk for ankle recurrent injury .

Recent studies have identified core and joint stabilization, stretching, strengthening, balance, mobilization, and flexibility exercises as a pivotal factor in preventing knee injuries in volleyball . In addition to these training programs, which help promote safer landing mechanics, training proper landing is also beneficial in injury prevention both for knee injuries and for ankle injuries.

Motor imagery (MI) is a contemporary method defined as a mental simulation of an action that is not actually performed . There are multiple brain areas, mostly motor areas, accepted to be involved in MI, but there is little evidence explaining the underlying mechanisms. Especially, the prefrontal cortex, involved in executive functions, is shown to be activated during MI tasks, but their interaction are not fully defined . MI has been described as a promising technique to facilitate the learning and improvement of motor skills in sports, education, and rehabilitation areas involving physical applications. Although the effectiveness of motor imagery in improving performance and learning new motor skills in sports is known, there is no research on its preventive role against injuries. The primary aim of this study was to investigate the effect of motor imagery on improving injury-causing factors related to jumps and falls in volleyball players. The secondary aim of this study was to investigate the effect of motor imagery on cortical functions.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 15 and 25,
* Not have an injury that affects the player's training program
* Play regularly for a professional team.

Exclusion Criteria:

* had lower extremity injury in the last two months
* who had been diagnosed with attention deficit hyperactivity disorder

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Kinematic Analysis | 12 weeks
  The flexion angles of the hip, knee, and dorsiflexion of the ankle during jumping and landing will evaluated with the 'Dartfish Analysis System' as degree.This software possesses simultaneous recording and measurement capabilities and is compatible with mobile phones for installation. This software is employed as a clinical instrument to measure movement amplitude and velocity, biaxial spatial coordinates, and joint angles throughout movement in the volleyball players

SECONDARY OUTCOMES:
Cognitive Functions | 12 weeks
  The Computerized Neurocognitive Tests Vital Sign (CNSVS) test consists of 10 standardized neurocognitive tests: verbal memory test, visual memory test, finger tapping test, symbol digit coding test, stroop test (simple reaction test, complex reaction test, and stroop effect), shifting attention test, continuous performance test, perception of emotions test, non-verbal reasoning test, and 4-part continuous performance test

CONTACTS AND LOCATIONS:
Locations (1):
- Fizyoostea, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Local regulations do not allow us to share participant information.

REFERENCES:
- [Background] Prasomsri J, Thueman B, Yuenyong P, Thongnoon C, Khophongphaibun N, Ariyawatcharin S. Effectiveness of motor imagery on sports performance in football players: A randomised control trial. Hong Kong Physiother J. 2024 Jun;44(1):29-37. doi: 10.1142/S1013702524500021. Epub 2023 Aug 25. PMID 38577393
- [Background] Deng N, Soh KG, Abdullah BB, Huang D. Does Motor Imagery Training Improve Service Performance in Tennis Players? A Systematic Review and Meta-Analysis. Behav Sci (Basel). 2024 Mar 5;14(3):207. doi: 10.3390/bs14030207. PMID 38540510
- [Background] Ridderinkhof KR, Brass M. How Kinesthetic Motor Imagery works: a predictive-processing theory of visualization in sports and motor expertise. J Physiol Paris. 2015 Feb-Jun;109(1-3):53-63. doi: 10.1016/j.jphysparis.2015.02.003. Epub 2015 Mar 25. PMID 25817985
- [Background] Kotegawa K, Teramoto W. Association of executive function capacity with gait motor imagery ability and PFC activity: An fNIRS study. Neurosci Lett. 2022 Jan 1;766:136350. doi: 10.1016/j.neulet.2021.136350. Epub 2021 Nov 13. PMID 34785311
- [Background] Zhang LL, Pi YL, Shen C, Zhu H, Li XP, Ni Z, Zhang J, Wu Y. Expertise-Level-Dependent Functionally Plastic Changes During Motor Imagery in Basketball Players. Neuroscience. 2018 Jun 1;380:78-89. doi: 10.1016/j.neuroscience.2018.03.050. Epub 2018 Apr 7. PMID 29634999
- [Background] Ruffino C, Papaxanthis C, Lebon F. Neural plasticity during motor learning with motor imagery practice: Review and perspectives. Neuroscience. 2017 Jan 26;341:61-78. doi: 10.1016/j.neuroscience.2016.11.023. Epub 2016 Nov 25. PMID 27890831
- [Background] Canepa P, Sbragi A, Saino F, Biggio M, Bove M, Bisio A. Thinking Before Doing: A Pilot Study on the Application of Motor Imagery as a Learning Method During Physical Education Lesson in High School. Front Sports Act Living. 2020 Oct 6;2:550744. doi: 10.3389/fspor.2020.550744. eCollection 2020. PMID 33345114
- [Background] Neilson V, Ward S, Hume P, Lewis G, McDaid A. Effects of augmented feedback on training jump landing tasks for ACL injury prevention: A systematic review and meta-analysis. Phys Ther Sport. 2019 Sep;39:126-135. doi: 10.1016/j.ptsp.2019.07.004. Epub 2019 Jul 19. PMID 31351340
- [Background] Ghaderi M, Letafatkar A, Thomas AC, Keyhani S. Effects of a neuromuscular training program using external focus attention cues in male athletes with anterior cruciate ligament reconstruction: a randomized clinical trial. BMC Sports Sci Med Rehabil. 2021 May 8;13(1):49. doi: 10.1186/s13102-021-00275-3. PMID 33964961
- [Background] Milic V, Radenkovic O, Capric I, Mekic R, Trajkovic N, Spirtovic O, Konicanin A, Bratic M, Mujanovic R, Preljevic A, Muric B, Kahrovic I. Sports Injuries in Basketball, Handball, and Volleyball Players: Systematic Review. Life (Basel). 2025 Mar 24;15(4):529. doi: 10.3390/life15040529. PMID 40283084
- [Background] Kilic O, Maas M, Verhagen E, Zwerver J, Gouttebarge V. Incidence, aetiology and prevention of musculoskeletal injuries in volleyball: A systematic review of the literature. Eur J Sport Sci. 2017 Jul;17(6):765-793. doi: 10.1080/17461391.2017.1306114. Epub 2017 Apr 9. PMID 28391750
- [Background] Wu CK, Lin YC, Lai CP, Wang HP, Hsieh TH. Dynamic Taping Improves Landing Biomechanics in Young Volleyball Athletes. Int J Environ Res Public Health. 2022 Oct 21;19(20):13716. doi: 10.3390/ijerph192013716. PMID 36294294
- [Background] McGuine TA, Post EG, Biese KM, Kliethermes S, Bell DR, Watson AM, Brooks A, Lang PJ. Incidence and Risk Factors for Injuries in Girls' High School Volleyball: A Study of 2072 Players. J Athl Train. 2023 Feb;58(2):177-184. doi: 10.4085/182-20. Epub 2020 Nov 5. PMID 33150377
- [Background] Skazalski C, Whiteley R, Sattler T, Kozamernik T, Bahr R. Knee, Low Back, and Shoulder Problems Among University and Professional Volleyball Players: Playing With Pain. J Athl Train. 2024 Jan 1;59(1):81-89. doi: 10.4085/1062-6050-0476.22. PMID 36913632
- [Background] Reeser JC, Gregory A, Berg RL, Comstock RD. A Comparison of Women's Collegiate and Girls' High School Volleyball Injury Data Collected Prospectively Over a 4-Year Period. Sports Health. 2015 Nov-Dec;7(6):504-10. doi: 10.1177/1941738115600143. Epub 2015 Aug 10. PMID 26502443